CLINICAL TRIAL: NCT07305545
Title: Investigation of the Effect of Massage Therapy on Sleep Duration and Mother-Baby Bonding in 0-6 Month Term Infants
Brief Title: Investigation of the Effect of Massage Therapy on Sleep Duration and Mother-Baby Bonding in Newborn
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, GÖZDE ARICA, research assisstant, University of Yalova
Other Study IDs: 2024/2
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Massage; Sleep; Newborn
MeSH Terms: interventions — Massage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interventional group: Group to be applied baby massage
  Interventions: Other: massage
- non-intervention group: Group not to be applied baby massage

INTERVENTIONS:
Other: massage — Basic classical baby massage, which is also taught to physiotherapists as part of their training. Classical massage will be applied to the baby's entire body, including the face.
  Groups: Interventional group

SUMMARY:
As the role of mothers increases in the postpartum period, depression, stress, sleep problems and general needs also increase. Recent studies have emphasized the need to treat more than just the mother's depression in cases of postpartum depression. The increase in the bond with the baby during this process is possible with the mother's compliance with the process. A healthy sleep between the mother and the baby improves the bond between them. One of the most important aids that facilitates the meeting of this need is baby massage. Baby massage is a tradition that begins immediately after birth in many cultures. Massage has a great positive effect on mother-baby interaction, increases the baby's sleep quality, reduces crying, lowers bilirubin levels and encourages mother-baby interaction. The aim of this study is to examine the effect of baby massage therapy applied by a physiotherapist on the baby's sleep duration and mother-baby attachment and the relationship between sleep duration and mother-baby attachment. The hypothesis of the study is that massage applied to babies will increase the baby's sleep quality and strengthen the bond between mother and baby.

ELIGIBILITY:
Inclusion Criteria:

* to be born on time
* to be between 0-6 months old

Exclusion Criteria:

* Conditions contraindicated for massage
* Termination of volunteering by guardian

Ages: 0 Days to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy babies, aged 0-6 months and born at term, whose parents' consent has been obtained will be included in the study.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Brief Infant Sleep Questionnaire | 4 weeks
  This questionnaire asks everything you need to know about baby sleep.
mother infant attachment scale | 4 weeks
  This scale is answered by the mother. It measures the mother's level of bonding with her baby.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Yalova, Yalova, Center, Turkey (Türkiye)